CLINICAL TRIAL: NCT05358223
Title: Comparison of the Effects of Music and Tens Application on Patient's Perception on Pain and Anxiety During Transrectal Prostate Biopsy
Brief Title: Pain and Anxiety During Transrectal Prostate Biopsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Reha Girgin, Assist.Prof.Dr.., Zonguldak Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: OR-9374
Record Dates: First submitted 2022-04-21; First posted 2022-05-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Prostate Biopsy
Keywords: pain; periprostatic block; transcutaneous electrical stimulation; music
MeSH Terms: conditions — Pain | interventions — Music Therapy; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Intervention Model Description: Patients who applied to the urology outpatient clinic and whose prostate biopsy decision was made according to the criteria specified in the guidelines of the European Urology Society, firstly detailed information about the study will be given after excluding those who were not suitable for the study, and then they will be randomly divided into 5 groups with the help of a computer program.
Masking Description: Due to the design of the study, it is not possible for patients and specialists to be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Prostatic block (No Intervention): Patients who will be treated with periprostatic block
- Prostatic block+Music (Active Comparator): Patients who will be treated with periprostatic block and who will be simultaneously listened to music
  Interventions: Other: Music
- Prostatic block+Tens (Active Comparator): Patients who will undergo periprostatic block and concomitant TENS
  Interventions: Device: TENS
- Music (Active Comparator): Patients who will only listen to music without periprostatic block
  Interventions: Other: Music
- Tens (Active Comparator): Patients who will only be treated with TENS without periprostatic block
  Interventions: Device: TENS

INTERVENTIONS:
Other: Music — A standard music determined by us for the 1st and 4th groups will be played during the process.
  Arms: Music; Prostatic block+Music
Device: TENS — TENS device will be connected to the 3rd and 5th groups during the process and the process will be done in this way.
  Arms: Prostatic block+Tens; Tens

SUMMARY:
Many studies have been conducted in the literature to manage pain and anxiety levels for patients undergoing transrectal prostate biopsy. In addition to the periprostatic block application recommended in the guidelines of the European Association of Urology, there are studies showing that TENS application or music applications will make an additional contribution.However, there is no study comparing the effect of TENS and music.

DETAILED DESCRIPTION:
Patients who applied to the urology outpatient clinic and whose prostate biopsy decision was made in accordance with the criteria specified in the guidelines of the European urology society will be randomized into 5 groups.

group 1: will apply only periprostatic block group 2: patients who will undergo periprostatic block + listen to music group 3 : patients to whom periprostatic block will be applied + tens device will be applied group 4 : patients who will only listen to music group 5 : patients who will only be treated with tens

A standard music determined by us for the 1st and 4th groups will be played during the process.

TENS device will be connected to the 3rd and 5th groups during the process and the process will be done in this way.

In our study, a 2-channel TENS device will be used. One of the electrodes connected to the first channel will be placed in the right anterior suprapubic region and the other in the right posterior presacral area. The electrodes connected to the second channel will be placed in the left anterior suprapubic region and left posterior presacral region, similar to the other. At least 3-6 minutes before the biopsy, stimulation will be started from the lower energy rising to 60 milliamperes with a frequency of 100 Hz and a pulse width of 150 µs. the amplitude will be adjusted individually for each participant to a level they can tolerate.

The blood pressure, pulse, respiratory rate and spo2 values of the patients are measured at the beginning, middle and end of the procedure and recorded. In our study, these data will be used by obtaining from the files of the patients.

In all groups, at the beginning, middle and end of the prostate biopsy procedure, an evaluation will be made with a visual analog score to evaluate the pain status of the patients.

Anxiety levels will be calculated with the state-continuity and anxiety scale that will be given to the patients the day before the procedure in all groups. After the prostate biopsy procedure is completed, this scale will be given to the patients again and their anxiety status will be re-evaluated after the procedure.

All the obtained data will be compared between these five groups and it will be tried to determine the optimal method in the pain and anxiety management of the patients.

Parameters to be used in the research:

* total psa , free psa , hemogram , urea, creatinine, total testosterone.
* International prostate symptom score ( IPSS ) and international erectile function index (IIEF- 5) score of 5 questions
* Visual analog pain score and state-continuity and anxiety scale scale
* Patients' blood pressure, fever, pulse and spo2 values

ELIGIBILITY:
Inclusion Criteria:

* Patients over 50 with high psa
* Patients with a family history of psa elevation over the age of 45
* psa > 10 ng/ml
* Patients with abnormal prostate examination
* Patients with psa 4-10 who need prostate biopsy
* Presence of PIRAD-4 and 5 lesions in multiparametric MR imaging
* Patients with consent to participate in the study

Exclusion Criteria:

* Patients with acute prostatitis
* Neutropenic patients
* Patients with bleeding diathesis that interferes with the procedure
* Patients without consent to participate in the study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2023-03-14 (Estimated); Study Completion 2023-03-14 (Estimated)

PRIMARY OUTCOMES:
pain during procedure | during the procedure
  VAS (visual analog scale) will be used for pain evaluation. A scale rating from 0 (no pain) to 10 (most painful).

SECONDARY OUTCOMES:
anxiety related to procedure | during the procedure
  STAI (The State-Trait Anxiety Inventory) will be used for anxiety evaluation. The STAI consists of 40 items, 20 for each subscale. Items are rated on a Likert scale from 1 (not at all/almost never) to 4 (very much so/almost always), and some items are reverse-scored.

CONTACTS AND LOCATIONS:
Overall Officials: Reha GİRGİN, Assist.Prof., Study Director — Zonguldak Bulent Ecevit University
Locations (1):
- Zonguldak Bulent Ecevit University, Zonguldak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No